CLINICAL TRIAL: NCT03800693
Title: Phase II Evaluation of the Effect of 2 Versus 6 Hour Oxaliplatin Infusions on Neuropathy and Pharmacokinetics in Patients With Gastrointestinal Cancers
Brief Title: 2 Versus 6 Hour Oxaliplatin Infusions in Patients With Gastrointestinal Cancers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Hematology/Oncology Pharmacy Association (Unknown); University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Olumide Gbolahan, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00106610; NCI-2018-02241 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship4468-18 (Other: Emory University Hospital/Winship Cancer Institute)
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Malignant Digestive System Neoplasm
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Fluorouracil; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 2-hour infusion group (Active Comparator): Patients receive oxaliplatin IV and leucovorin IV over 2 hours on day 1. Patients also receive a lower dose of fluorouracil IV over 2-4 minutes followed by a higher dose IV continuous over 4-6 hours on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin
- 6-hour infusion group (Experimental): Patients receive oxaliplatin IV over 6 hours on day 1. Patients also receive leucovorin and fluorouracil as in the 2-hour infusion group. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Fluorouracil — Given IV
  Other Names: 5-FU; Carac; Ribofluor
Drug: Leucovorin — Given IV
  Other Names: Folinic acid
Drug: Oxaliplatin — Given IV
  Other Names: Eloxatin

SUMMARY:
This phase II trial studies how well giving oxaliplatin over 6 hours works in treating nerve damage in patients with gastrointestinal cancers. Oxaliplatin can cause side effects such as nerve damage that may delay or reduce the dose of oxaliplatin. Giving oxaliplatin over a longer period of time (6 hours) may prevent or delay the development of nerve damage, which may keep patients on standard doses of chemotherapy longer, without having to delay treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the effect of 2 versus 6-hour oxaliplatin infusion time on the difference in severity of sensory neuropathy as measured by patient reported outcome (PRO) scores on the European Organization for Research and Treatment of Cancer (EORTC) chemotherapy-induced peripheral neuropathy (CIPN-20) scale at the initiation of cycle 4.

SECONDARY OBJECTIVES:

I. Pharmacokinetic parameters of maximum concentration (Cmax), area under the curve (AUC), time of maximum concentration (tmax), clearance, and half life (t1/2) of platinum ultra-filtrate.

II. CIPN-20 sensory score changes over the duration of therapy as measured by a cumulative area-under-the curve score.

III. Clinical outcomes including duration of therapy, oxaliplatin dose reductions, delays in therapy, and overall dose intensity and delivery of oxaliplatin.

IV. Relationship between oxaliplatin Cmax, patient-reported acute neurotoxicity, and chronic neurotoxicity by CIPN-20 scores.

OUTLINE: Patients are randomized to 1 of 2 groups.

2-hour infusion group: Patients receive oxaliplatin intravenously (IV) and leucovorin IV over 2 hours on day 1. Patients also receive a lower dose of fluorouracil IV over 2-4 minutes followed by a higher dose IV continuous over 4-6 hours on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

6-hour infusion group: Patients receive oxaliplatin IV over 6 hours on day 1. Patients also receive leucovorin and fluorouracil as in the 2-hour infusion group. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 1, 3, 6, 12, and 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Confirmed diagnosis of a gastrointestinal cancer
* Plan for 4 or more cycles of FOLFOX6 (fluorouracil [with leucovorin] and oxaliplatin) containing chemotherapy
* Histologically confirmed, measurable or evaluable disease. Patients with advanced or metastatic disease should have at least one measurable lesion by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Patients in the adjuvant treatment setting planned to have > 4 cycles of FOLFOX-containing chemotherapy are eligible and will be followed per standard of care
* Absolute neutrophil count (ANC) ≥ 1,500/µL (no white blood cell growth factors allowed to meet requirement)
* Platelets ≥ 75,000/µL (may be transfused up to 72 hours prior to day 1 to meet requirement)
* Hemoglobin ≥ 8 g/dL (may be transfused up to 72 hours prior to day 1 to meet requirement)
* Creatinine clearance > 30 mL/min by Cockcroft-Gault, to preserve similar dosing (85 mg/m²) for analysis
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
* Signed informed consent
* Adequate birth control when appropriate

Exclusion Criteria:

* Any preexisting grade 2 or higher peripheral neuropathy
* Patients currently receiving anticancer therapies or who have received any focal or systemic anticancer therapy within 14days of the start of FOLFOX6
* Known intolerance or hypersensitivity to any agent in FOLFOX6 or concurrent agents
* Patients who have any known severe and/or uncontrolled medical conditions such as:

  * Unstable angina pectoris, symptomatic heart failure; (New York Heart Association class III or IV), myocardial infarction ≤ 6 months prior, serious uncontrolled cardiac arrhythmia, or any other clinically significant cardiac disease
  * Active (acute or chronic) or uncontrolled severe infection, liver disease such as cirrhosis, or decompensated liver disease
* Patients with any history of severe hemorrhage requiring ≥ 4 units of packed red blood cells (RBCs) in a 48-hour period
* Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will not be able to complete the entire study
* Patients who are currently part of or have participated in any clinical investigation with an investigational drug within 14days prior to dosing
* Pregnant or nursing (lactating) women
* Women of childbearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, must use highly effective methods of contraception during the study and 8 weeks after. Highly effective contraception methods include combination of any two of the following:

  * Use of oral, injected or implanted hormonal methods of contraception or;
  * Placement of an intrauterine device (IUD) or intrauterine system (IUS);
  * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository;
  * Total abstinence or;
  * Male/female sterilization Women are considered post-menopausal and not of childbearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks prior to randomization. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of childbearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-03-14 (Actual); Primary Completion 2026-08-05 (Estimated); Study Completion 2026-09-17 (Estimated)

PRIMARY OUTCOMES:
Effect of 2 versus 6-hour oxaliplatin infusion time on neuropathy as measured by patient reported outcome (PRO) scores on the European Organization for Research and Treatment of Cancer (EORTC) chemotherapy-induced peripheral neuropathy (CIPN-20) scale | Baseline up to 60 days (course 4)
  The EORTC-CIPN-20 sub-scales will be computed according to the standard scoring algorithm and then transformed to a 0 to 100 scale, where high scores mean less symptom burden. The primary outcome measure of difference in sensory scores of the two groups between baseline and the initiation of cycle 4 will be the driver of the analysis.

SECONDARY OUTCOMES:
Maximum concentrations achieved (Cmax) | At baseline and at 1, 2, 4, 6, 48, and 192 hours after initiation of oxaliplatin
  The study will focus on maximum concentrations achieved (Cmax) with each infusion time. Data will be analyzed using non-compartmental methods via Phoenix WinNonlin analytical software, version 8.0 or higher.
Changes in tumor size | Up to 18 months after completion or discontinuation of chemotherapy
  The study will assess changes in tumor size per standard of care assessments at screening and every 2 months.
Duration of therapy | Up to 18 months after completion or discontinuation of chemotherapy
  Duration of therapy will be recorded.
Dose density | Up to 18 months after completion or discontinuation of chemotherapy
  Dose density will be recorded.
Frequency of dose holds or reductions | Up to 18 months after completion or discontinuation of chemotherapy
  Frequency of dose holds or reductions will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Olumide B. Gbolahan, MBBS, MSc, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No